CLINICAL TRIAL: NCT01515176
Title: Phase 1b/2 Study of Dinaciclib (SCH 727965) and Ofatumumab in Relapsed and Refractory CLL/SLL/B-PLL
Brief Title: Ofatumumab and Dinaciclib in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia, Small Lymphocytic Lymphoma, or B-Cell Prolymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00101; NCI-2012-00101 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-11120; OSU11120; CDR0000721353; OSU 11120 (Other: Ohio State University Comprehensive Cancer Center); 9031 (Other: CTEP); N01CM00070 (NIH); N01CM62207 (NIH); P30CA016058 (NIH); P50CA140158 (NIH); U01CA076576 (NIH); UM1CA186712 (NIH)
Record Dates: First submitted 2012-01-16; First posted 2012-01-23 (Estimated); Results first posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-02

CONDITIONS: Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic | interventions — dinaciclib; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ofatumumab, dinaciclib) (Experimental): Patients receive ofatumumab IV over 4-6 hours on days 1, 8, 15, and 22 of courses 1-2, and on day 1 of courses 4-7. Beginning on course 2, patients also receive dinaciclib IV over 2 hours on days 2, 8, and 15 of course 2, and on days 1, 8, and 15 of courses 3-7. Treatment repeats every 28 days for up to 7 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dinaciclib; Other: Laboratory Biomarker Analysis; Biological: Ofatumumab; Other: Pharmacological Study

INTERVENTIONS:
Drug: Dinaciclib — Given IV
  Other Names: CDK Inhibitor SCH 727965; MK-7965; SCH 727965
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Ofatumumab — Given IV
  Other Names: Arzerra; GSK1841157; HuMax-CD20; HuMax-CD20, 2F2
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and the best dose of ofatumumab and dinaciclib and to see how well they work in treating patients with relapsed or refractory chronic lymphocytic leukemia, small lymphocytic lymphoma, or B-cell prolymphocytic leukemia. Monoclonal antibodies, such as ofatumumab, can find cancer cells and help kill them. Dinaciclib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving ofatumumab together with dinaciclib may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the tolerable dose of combination therapy with ofatumumab and dinaciclib (phase 1b component) in chronic lymphocytic leukemia (CLL), small lymphocytic leukemia (SLL), and B-cell prolymphocytic leukemia (B-PLL).

II. To characterize the toxicity of combination therapy with ofatumumab and dinaciclib in CLL/SLL/B-PLL.

III. To determine the overall response rate associated with this treatment as assessed by consensus response criteria. (Phase II)

SECONDARY OBJECTIVES:

I. To estimate progression-free survival (PFS) after combination treatment with ofatumumab and dinaciclib.

II. To characterize the pharmacokinetics of dinaciclib when given in combination with ofatumumab.

III. To correlate pharmacokinetic features of dinaciclib with response, toxicity (particularly tumor lysis syndrome), and pharmacodynamic endpoints.

IV. To perform detailed baseline and serial pharmacodynamic studies of combination therapy with ofatumumab and dinaciclib and correlate these with response to therapy.

V. To correlate baseline disease-risk parameters (i.e., zeta-chain-associated protein kinase [ZAP]-70 expression, interphase cytogenetics, immunoglobulin heavy chain variable region [IgVH] mutational analysis, and other clinical prognostic factors) with response to therapy.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive ofatumumab intravenously (IV) over 4-6 hours on days 1, 8, 15, and 22 of courses 1-2, and on day 1 of courses 4-7. Beginning on course 2, patients also receive dinaciclib IV over 2 hours on days 2, 8, and 15 of course 2, and on days 1, 8, and 15 of courses 3-7. Treatment repeats every 28 days for up to 7 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed B-cell chronic lymphocytic leukemia (B-CLL)/small lymphocytic lymphoma (SLL) or a B-cell prolymphocytic leukemia (B-PLL) according to 2008 World Health Organization (WHO) diagnostic criteria
* Patients must meet one or more of the following modified indications for treatment as described in the 2008 International Workshop on chronic lymphocytic leukemia (CLL) (IWCLL) guidelines for the diagnosis and treatment of CLL:

  * Progressive disease or marked splenomegaly and/or lymphadenopathy or disease requiring de-bulking for future allogeneic transplantation
  * Anemia (hemoglobin < 11 mg/dL) or thrombocytopenia (platelets < 100,000/μL)
  * Unexplained weight loss exceeding 10% of body weight over the preceding 6 months
  * Cancer Therapy Evaluation Program (CTEP) active version of the Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or 3 fatigue
  * Fevers > 100.5 º F or night sweats for greater than 2 weeks without evidence of infection
  * Progressive lymphocytosis, with an increase exceeding 50% over a 2-month period or a doubling time of less than 6 months
  * Need for cytoreduction prior to allogeneic stem cell transplant
* Patients must have received at least one prior therapy that includes either fludarabine or equivalent nucleoside analogue, or an alternative regimen if there was a contraindication (i.e. autoimmune hemolytic anemia) or patient elected not to receive fludarabine
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy >= 12 weeks
* Absolute neutrophil count >= 1,000/μL in absence of bone marrow involvement
* Platelets >= 30,000/μL in absence of bone marrow involvement
* Total bilirubin =< 1.5 X institutional upper limit of normal (ULN) unless secondary to Gilbert's
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal (ULN) unless due to infiltration of the liver
* Creatinine =< 2.0 mg/dL OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients(Cockcroft-Gault estimated)
* Patients with a history of current/previous infection with hepatitis B virus will be eligible if receiving appropriate antiviral prophylaxis
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier; corticosteroids alone will not be considered prior therapy, but must be discontinued at least 24 hours prior to the first day of therapy unless continued for indications other than the primary malignancy
* Patients who are receiving any other investigational agents
* Patients who have received prior treatment with dinaciclib will not be eligible; patients previously treated with ofatumumab will be eligible as long as their disease responded to previous treatment (defined as achieving at least stable disease by consensus criteria) and did not subsequently progress < 3 months from completing treatment
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition as dinaciclib
* History of anaphylactic reaction to rituximab or other anti-cluster of differentiation (CD)20 monoclonal antibody
* Because dinaciclib is metabolized by the cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) liver enzyme, the eligibility of patients taking medications that are potent inducers or inhibitors of that enzyme will be determined following a review of their case by the principal investigator; every effort should be made to switch patients taking such agents or substances to other medications; any identified agent needs to be stopped at least 2 weeks prior to study registration; use of aprepitant will be permitted, however, based on drug-drug interaction study performed by the manufacturer showing no effect on dinaciclib pharmacokinetics (PK)
* Patients with glucose-6-phosphate dehydrogenase (G6PD) deficiency are excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and/or breast-feeding women are excluded from this study; breastfeeding should be discontinued if the mother is treated with dinaciclib
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject is considered by his or her physician to have a 2 year survival expectation
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-03-04 (Actual); Study Completion 2016-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Rogers, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level I: Treatment (Ofatumumab, Dinaciclib): Patients receive ofatumumab IV over 4-6 hours on days 1, 8, 15, and 22 of courses 1-2, and on day 1 of courses 4-7. Beginning on course 2, patients also receive dinaciclib 7 mg/m2 as a 2-hour infusion on cycle 2 day 2, escalated to 10 mg/m2 beginning with cycle 2 day 8 and continuing thereafter.
- Dose Level II: Treatment (Ofatumumab, Dinaciclib): Patients receive ofatumumab IV over 4-6 hours on days 1, 8, 15, and 22 of courses 1-2, and on day 1 of courses 4-7. Beginning on course 2, patients also receive dinaciclib 7 mg/m2 as a 2-hour infusion on cycle 2 day 2, escalated to 10 mg/m2 as a 2-hour infusion on cycle 2 day 8, and to 14 mg/m2 on cycle 2 day 15 and continuing thereafter
Period: Overall Study
Arm/Group | Dose Level I: Treatment (Ofatumumab, Dinaciclib) | Dose Level II: Treatment (Ofatumumab, Dinaciclib)
Started | 4 | 32
Completed | 4 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level II:: Patients receive ofatumumab IV over 4-6 hours on days 1, 8, 15, and 22 of courses 1-2, and on day 1 of courses 4-7. Beginning on course 2, patients also receive dinaciclib 7 mg/m2 as a 2-hour infusion on cycle 2 day 2, escalated to 10 mg/m2 as a 2-hour infusion on cycle 2 day 8, and to 14 mg/m2 on cycle 2 day 15 and continuing thereafter
- Total: Total of all reporting groups
Arm/Group | Dose Level I: Treatment (Ofatumumab, Dinaciclib) | Dose Level II: | Total
Number analyzed (Participants) | 4 | 32 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 15 | 17
  >=65 years | 2 | 17 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 11 | 13
  Male | 2 | 21 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 32 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 4 | 27 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 32 | 36

OUTCOME MEASURES:

1. Primary Outcome: Maximum-tolerated Dose of Dinaciclib When Given in Combination With Ofatumumab, Defined as a Dose Level Where at Most One of 6 Evaluable Patients Has a Dose Limiting Toxicity (Phase Ia)
Description: Graded according to the National Cancer Institute (NCI) CTCAE version (v)4.0. Assessed using the continuous variables as the outcome measures (primarily nadir and percent change from baseline values) as well as categorization.
Time Frame: Day 56
Measure: Number; unit: mg/m2
Arm/Group | Treatment (Ofatumumab, Dinaciclib)
Number analyzed (Participants) | 36
mg/m2
  2 hr infusion cycle 2 day 2 | 7
  2 hr infusion cycle 2 day 8 | 10
  cycle 2 day 8 | 14

2. Primary Outcome: Number of Patients With Dose-limiting Toxicity Incidents Graded According to the NCI CTCAE v4.0 (Phase I)
Description: Hematologic dose-limiting toxicity measures will be assessed using the continuous variables as the outcome measures (primarily nadir and percent change from baseline values) as well as categorization via CTCAE version 4 standard toxicity grading. Non-hematologic dose-limiting toxicities such as dyspnea and renal will be evaluated via the ordinal CTCAE standard toxicity grading only.
Time Frame: Up to day 56
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level I: Treatment (Ofatumumab, Dinaciclib) | Dose Level II: Treatment (Ofatumumab, Dinaciclib)
Number analyzed (Participants) | 4 | 32
Participants | 0 | 0

3. Primary Outcome: Percentage of Patients Who Achieve an Overall Response, Defined as Achieving a Complete Response, an Unconfirmed Complete Response (SLL Only), or a Partial Response (Phase II)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 28 weeks
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Dose Level I and Dose Level II: Dose Level I:
  Patients receive ofatumumab IV over 4-6 hours on days 1, 8, 15, and 22 of courses 1-2, and on day 1 of courses 4-7.
  Dose Level II:
  Patients receive ofatumumab IV over 4-6 hours on days 1, 8, 15, and 22 of courses 1-2, and on day 1 of courses 4-7. Beginning on course 2, patients also receive dinaciclib IV over 2 hours on days 2, 8, and 15 of course 2, and on days 1, 8, and 15 of courses 3-7. Treatment repeats every 28 days for up to 7 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Dose Level I and Dose Level II
Number analyzed (Participants) | 36
percentage of patients | 39 [23 to 57]

4. Secondary Outcome: Complete Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions
Time Frame: Up to 28 weeks
Measure: Number (95% Confidence Interval); unit: patients with complete response
Arm/Group | Treatment (Ofatumumab, Dinaciclib)
Number analyzed (Participants) | 36
patients with complete response | 0 [0 to 0]

5. Secondary Outcome: Overall Survival
Description: Distributions will be explored and assessed using the methods of Kaplan and Meier.
Time Frame: Time from study entry to death due to any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Ofatumumab, Dinaciclib)
Number analyzed (Participants) | 36
days | 990 [678 to NA] — Time point to reach the lower bound of 95% CI for median survival rate not reached yet

6. Secondary Outcome: Progression Free Survival
Description: 95% confidence intervals will be constructed using the methods of Duffy and Santner with the assumption that these rates are binomially distributed. Distributions will be explored and assessed using the methods of Kaplan and Meier.
Time Frame: Time from study entry to documentation of disease progression and/or death, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dose Level I and Dose Level II
Number analyzed (Participants) | 36
days | 322 [223 to 402]

7. Secondary Outcome: Time to Treatment Failure
Description: Distributions will be explored and assessed using the methods of Kaplan and Meier.
Time Frame: Time from study entry to the date patients end treatment, up to 28 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Ofatumumab, Dinaciclib)
Number analyzed (Participants) | 36
days | 248 [113 to 347]

ADVERSE EVENTS:
Description: All toxicities will be assessed using the CTEP Active Version of the NCI Common Terminology Criteria for Adverse Events (CTCAE).
Arm/Group | Dose Level I: Treatment (Ofatumumab, Dinaciclib) | Dose Level II: Treatment (Ofatumumab, Dinaciclib)
All-Cause Mortality (participants affected / at risk) | 0/4 | 1/32
Serious Adverse Events (participants affected / at risk) | 3/4 | 32/32
Other Adverse Events (participants affected / at risk) | 4/4 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level I: Treatment (Ofatumumab, Dinaciclib) (N=4) | Dose Level II: Treatment (Ofatumumab, Dinaciclib) (N=32)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HEART FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1)
DEATH NOS (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 2 (3)
CATHETER RELATED INFECTION (Infections and infestations) | 0 (0) | 1 (1)
HEPATITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 4 (5)
PLEURAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 3 (3)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 1 (2)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 (0) | 12 (14)
TUMOR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HEMATOMA (Vascular disorders) | 0 (0) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level I: Treatment (Ofatumumab, Dinaciclib) (N=4) | Dose Level II: Treatment (Ofatumumab, Dinaciclib) (N=32)
Anemia (Blood and lymphatic system disorders) | 3 (7) | 28 (54)
Lymphode Pain (Blood and lymphatic system disorders) | 0 (0) | 6 (8)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 3 (5)
Constipation (Gastrointestinal disorders) | 1 (2) | 11 (15)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 12 (18)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 6 (7)
Mucositis (Gastrointestinal disorders) | 0 (0) | 4 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 10 (12)
Oral Dysesthesia (Gastrointestinal disorders) | 0 (0) | 3 (4)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (5)
Chills (General disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 2 (2) | 15 (18)
Fever (General disorders) | 1 (1) | 2 (2)
General Disorders and Administration site Conditions-other (General disorders) | 1 (1) | 0 (0)
Infusion Related Reactions (General disorders) | 0 (0) | 3 (3)
Pain (General disorders) | 3 (3) | 6 (6)
Lung Infection (Infections and infestations) | 0 (0) | 2 (3)
Skin Infection (Infections and infestations) | 0 (0) | 2 (4)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 3 (4)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 2 (5) | 9 (14)
Alkaline Phosphatase Increased (Investigations) | 0 (0) | 12 (28)
Aspartate Aminotransferase Increased (Investigations) | 2 (5) | 9 (24)
Blood Bilirubin Decreased (Investigations) | 1 (1) | 4 (6)
Creatinine Increased (Investigations) | 0 (0) | 11 (19)
Investigations-Other (Investigations) | 0 (0) | 2 (2)
Lymphocyte Count Decreased (Investigations) | 2 (5) | 20 (57)
Lymphocyte Count Increased (Investigations) | 2 (3) | 14 (21)
Neutrophil Count Decreased (Investigations) | 4 (10) | 26 (91)
Platelet Count Decreased (Investigations) | 4 (4) | 23 (48)
Weight Gain (Investigations) | 0 (0) | 2 (2)
Weight Loss (Investigations) | 0 (0) | 3 (3)
White Blood Cell Decreased (Investigations) | 2 (4) | 22 (87)
Hypercalcemia (Investigations) | 0 (0) | 5 (8)
Hyperglycemia (Investigations) | 4 (10) | 31 (84)
Hyperkalemia (Investigations) | 0 (0) | 8 (8)
Hypermagnesemia (Investigations) | 1 (1) | 2 (2)
Hypernatremia (Investigations) | 0 (0) | 3 (3)
Hyperuricemia (Investigations) | 0 (0) | 7 (10)
Hypoalbuminemia (Investigations) | 3 (5) | 19 (23)
Hypocalcemia (Investigations) | 3 (5) | 18 (37)
Hypoglycemia (Investigations) | 0 (0) | 6 (7)
Hypokalemia (Investigations) | 2 (3) | 17 (21)
Hypomagnesemia (Investigations) | 2 (3) | 7 (20)
Hyponatremia (Investigations) | 1 (2) | 11 (13)
Hypophosphatemia (Investigations) | 1 (2) | 24 (45)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (9)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neoplasms benign, Malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 5 (6)
Dysesthesia (Nervous system disorders) | 0 (0) | 10 (11)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 9 (9)
Paresthesia (Nervous system disorders) | 2 (2) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (5)
Restlessness (Psychiatric disorders) | 0 (0) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (3)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (8)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hyperhidrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (8)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 22 (45)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less